CLINICAL TRIAL: NCT03663998
Title: DNAVAC 001: A Phase 1 Open-labelled Trial to Optimise DNA Vaccination for Antibody Induction
Brief Title: Optimising DNA Vaccinations in Healthy Volunteers
Acronym: DNAVAC001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 14SM2306
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: HIV-1-infection
Keywords: Antibody; Antibody-dependent cell-mediated cytotoxicity; Investigational Medicinal Product; neutralizing antibody responses

STUDY DESIGN:
Intervention Model Description: Groups A-F will be recruited sequentially, groups G and H once the optimal dose for IM has been determined, and group I selecting the optimal doses for IM and ID form groups A-F for combined administration. This will represent a divided dose group across two different anatomical sites. Each group will receive four vaccinations (at 0, 4, 8 and 12 weeks). The choice of four vaccinations is based on the observation that antibody responses to DNA vaccination in mice plateau after the fourth vaccination, while in rabbits after the third. Hence it is unclear where they may plateau in humans.
Masking Description: There will be no blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- A (Active Comparator): CN54ENV IM EP 400 g
  Interventions: Biological: CN54ENV DNA
- B (Active Comparator): CN54ENV IM EP 1000 g
  Interventions: Biological: CN54ENV DNA
- C (Active Comparator): CN54ENV IM EP 4000 g
  Interventions: Biological: CN54ENV DNA
- D (Active Comparator): CN54ENV ID EP 600 g
  Interventions: Biological: CN54ENV DNA
- E (Active Comparator): CN54ENV ID EP 1200 g
  Interventions: Biological: CN54ENV DNA
- F (Active Comparator): CN54ENV ID EP 1800 g
  Interventions: Biological: CN54ENV DNA
- G (Active Comparator): CN54ENV IM1 EP
  + pIL-12 (500 g)
  Interventions: Biological: GENEVAX® IL-12 DNA
- H (Active Comparator): CN54ENV IM1 EP
  + pIL-12 (1500 g)
  Interventions: Biological: GENEVAX® IL-12 DNA
- I (Active Comparator): CN54ENV IM1 EP
  + ID2 EP
  Interventions: Biological: CN54ENV DNA

INTERVENTIONS:
Biological: CN54ENV DNA — CN54ENV DNA concentration 4 ± 0.7 mg/mL is formulated in 1 x PBS
  All administrations of CN54ENV will be by in vivo electroporation using the Ichor Medical Systems TriGrid Delivery System for intramuscular (TDS-IM) or intradermal use (TDS-ID) and will be delivered into the upper thigh(s).
  Arms: A; B; C; D; E; F; I
Biological: GENEVAX® IL-12 DNA — GENEVAX® IL-12 DNA, concentration 2 mg/mL with a fill volume of 1.0 mL (1.0 ± 0.1mL), is formulated in 30 mM citrate buffer.
  GENEVAX® IL-12 DNA is mixed with the CN54ENV DNA immediately prior to administration.
  Arms: G; H

SUMMARY:
This is a two part study to evaluate the immunogenicity and tolerability of DNA-C CN54ENV plasmid DNA (CN54ENV) administered with electroporation (EP), with and without DNA encoding recombinant interleukin-12 (GENEVAX® IL-12). Part 1 is exploratory and designed to select conditions capable of promoting enhanced B cell responses in a limited number of volunteers. Part 2 is dependent upon Part 1 and is designed to study the fine specificity of the B-cell immune responses to CN54ENV DNA in an expanded number of subjects. Data from both stages will be combined for safety and immunological analysis.

DETAILED DESCRIPTION:
It is generally accepted that globally effective HIV-1 vaccine will likely need to induce bnAbs against HIV-1. The proposed study is based on the recognition of the potential strategic importance of performing iterative small human studies to accelerate HIV-1 immunogen discovery, where DNA vaccines offer the fastest and most cost effective approach for rapid screening of multiple immunogens. This study aims to leverage DNA immunization as a platform to accelerate the discovery of HIV-1 immunogens capable of inducing bnAbs in humans.

To meet this aim this study seeks to apply recent state of the art technological advances in DNA vaccination and immune monitoring, both at the single cell and molecular level, to enable detailed probing of developing vaccine induced antibody responses. In this respect it represents the first attempt in humans to use a DNA vaccine approach to investigate the development and focusing of B cell responses to vaccination. Should this approach be successful it will provide an important new strategy for rapidly conducting systematic clinical research studies in humans aimed at moving the HIV-1 vaccine field closer to achieving the key objective of identification of immunogens and vaccine strategies required for induction of bnAbs in humans.

At the end of 2012, an estimated 35.3 million people were living with HIV worldwide, up 17% from 2001. This reflects the continued large number of new HIV infections and a significant expansion of access to antiretroviral therapy, which has helped reduce AIDS-related deaths, especially in more recent years (UNAIDS Report on the global AIDS epidemic 2013. Geneva 2013). The majority of new HIV infections continue to occur in sub-Saharan Africa. There is an urgent need to strengthen and scale-up existing and new prevention methods such as HIV testing and counselling, behavioural interventions, condom use, treatment of sexually transmitted diseases, harm reduction, male circumcision (Wamai, Morris et al. 2011) and antiretroviral drugs for prevention (Granich, Gupta et al. 2011). New prevention strategies to control the epidemic and prevent new infections, including pre-exposure prophylaxis (Kim, Becker et al. 2010), antiviral treatment for prevention (Granich, Lo et al. 2011), topical microbicides (Krakower and Mayer 2011), and HIV preventive vaccines must be explored and their access ensured. However the development of an efficacious preventive vaccine against HIV-1 remains among the best hopes for controlling the HIV/AIDS pandemic (Kim, Rerks-Ngarm et al. 2010, Koff 2010).

Data from a recent community-based efficacy trial in Thailand (RV144) testing a vaccination regimen consisting of priming with the canarypox vector ALVAC-HIV, expressing HIV gag, pro, and env genes, and boosting with recombinant AIDSVAX B/E HIV Env protein demonstrated modest vaccine protection against HIV acquisition. The vaccine efficacy decreased over the first year after vaccination from 60% at one year to 31.2 % at 3.5 years post first vaccination, suggesting that protection may be related to HIV-specific antibodies waning over time (Rerks-Ngarm, Pitisuttithum et al. 2009). The regimen did not decrease HIV viral load in vaccine recipients who acquired HIV. CD8 T-cell responses were in few vaccine recipients, while binding antibodies were detected in a majority of them, with very limited detectable neutralizing antibody responses to HIV. These results suggest that more potent vaccines are needed for providing significant and sustained protection against HIV acquisition as well as for controlling viral replication.

Neutralizing antibodies against circulating isolates are induced principally by HIV Env and could potentially confer sterilizing immunity against HIV, as suggested by non-human primate SHIV challenge studies (Mascola, Stiegler et al. 2000, Pantophlet and Burton 2006, Hessell, Poignard et al. 2009). Moreover, a recent Non Human Primates (NHP) study demonstrates that SIV (Simian Immunodeficiency Virus) Env antigen was essential to confer protection against SIV challenge and that SIV Env-specific binding non-neutralizing antibodies played a role in this protection (Barouch, Liu et al. 2012). Previous trials using monomeric AIDSVAX gp120 showed no efﬁcacy in a phase III trials (Flynn, Forthal et al. 2005, Pitisuttithum, Gilbert et al. 2006). This failure has been a major drawback for Env-based HIV vaccines, since current immunogens afford only very narrow protection against HIV strains that are closely related to the vaccine antigen (Zhang and Dimitrov 2007, Montero, van Houten et al. 2008). In RV144, an analysis of the correlates of risk showed that IgG3 binding antibodies to scaffolded-V1V2 recombinant protein correlated inversely with infection rate while Env binding plasma IgA correlated directly with infection rate (Haynes, Gilbert et al. 2012). Several lines of evidence suggest that vaccine induced antibodies recognize conformational epitopes in the scaffolded V1V2 reagent, which has been shown to detect conformational V1V2 antibodies (Pinter, Honnen et al. 1998, Zolla-Pazner, deCamp et al. 2013). The results of an analysis of breakthrough viruses from patients in the RV144 trial were consistent with immune pressure focused on amino acid patterns in and flanking the V1V2 region of HIV-1 Env (Edlefsen, Gilbert et al. 2013). This region serves critical functions, such as participating in CD4-receptor and chemokine-receptor binding, binding to α4β7 integrin (Nawaz, Cicala et al. 2011) and serving as the binding site of neutralizing antibodies (Gorny, Stamatatos et al. 2005, Walker, Phogat et al. 2009, Changela, Wu et al. 2011, McLellan, Pancera et al. 2011). However, the search for an immunogen able to induce broad cross-protective and long-lasting neutralizing/functional antibodies remains difficult and critical (Burton, Desrosiers et al. 2004, Montefiori, Sattentau et al. 2007).

During the vast majority of natural HIV infections, the antibody response which develops is "too little, too late" - occurring approximately 12 weeks from initial exposure which is after viral expansion has occurred (McMichael, Borrow et al. 2010). Recent data also suggests that under normal circumstances, heterosexual transmission is a relatively rare event and that there is a small "window of opportunity" - in the order of days - during which it might be possible to stop the establishment of a latent infection. An ideal vaccine would prime a very early and broad antibody response targeting multiple neutralizing epitopes for effective control of early viral replication. However, bnAbs typically only arise in only 1% of chronically infected subjects, take several years to develop, display exceptional levels of somatic hyper mutation, have unusually long CDR3 regions and exhibit significant glycan-binding, properties not induced by current vaccine candidates. Thus elicitation of broadly neutralizing antibodies (bnAbs) against HIV-1 is both a problem of Immunogen Design and Human Immune Responsiveness.

Despite significant progress in identifying broadly neutralizing antibodies in a very small number of infected individuals, and detailed characterization of their cognate epitopes, attempts to design appropriate immunogens inducing HIV-specific broadly neutralizing antibodies have so far failed. Indeed, next generation vaccines are likely to be critically dependent upon discovery of novel immunogens capable of eliciting protective responses in humans. However, this is limited by the current lack of understanding as to how immunogens induce protective antibody responses, their gene usage, their maturation pathways, and factors facilitating breadth and potency. While animal studies have played an important role in understanding the pathogenesis of HIV and related retroviruses, they are quite limited when it comes to modelling human immunization studies due to differences in immunogenetics and species specificity. The advent of technological advances that probe human immune responsiveness at the single cell and molecular level now provide the necessary tools to look beyond pre-clinical models to resolve these issues. Indeed, a strong argument for increased and improved early clinical studies in humans (instead of the currently lengthy process of prior extensive animal testing) is that animals, including non-human primates (NHP), may not accurately recapitulate germline engagement of B cells, which could be critical for vaccines designed to induce HIV-1 envelope (Env) bnAbs. To resolve this, it is now generally agreed that rapid, iterative, small, experimental early human vaccine studies are needed to select and refine the best approaches to immunogen design. Such an approach would allow rapid selection of the most promising vaccine strategies at an early stage thereby reducing the risk of failure in more advanced phase clinical development. However, the cost and lengthy time lines associated with the manufacture of recombinant proteins means it is not feasible to test multiple iterations of HIV-1 envelope structures. In contrast, DNA vaccines offer a rapid and feasible approach for screening multiple immunogens in human trials based on ease of manufacture and reduced costs.

Although early approaches to DNA vaccination failed to induce significant antibody responses in humans, more recent trials have shown that DNA vaccines can induce neutralizing antibodies against a number of viruses (Martin, Pierson et al. 2007, Martin, Louder et al. 2008, Ledgerwood, Pierson et al. 2011, Ledgerwood, Hu et al. 2012) and detectable antibody responses to HIV-1 (Catanzaro, Roederer et al. 2007). Various strategies can now be used to improve and augment the immunogenicity of DNA vaccines including: promoter selection and codon optimization; the use of electroporation (EP); the route of administration (intramuscular (IM) or intradermal (ID)); and the use of molecular adjuvants such as IL-12 (Sardesai and Weiner 2011, Yin, Dai et al. 2011, Kopycinski, Cheeseman et al. 2012). The additional advantage provided by lack of anti-vector immunity associated with other delivery platforms (viral vectors) provides the opportunity for serial immunizations with multiple DNA derived immunogens. In this context DNA vaccination offers the potential to provide targeted germline priming that may critically redirect antibody responses upon protein boosting (Schittek and Rajewsky 1990, Yoshida, Mei et al. 2010). Furthermore, the lack of vector immunity would allow the use of a series of DNA encoded immunogens to engage germline B cells and direct them towards recognition of bnAb epitopes prior to amplification by protein boosting. While multiple dose DNA vaccination may not represent a practical approach to a prophylactic mass vaccination campaign, its potential to induce antibody responsiveness may make it an important clinical research tool for immunogen discovery and refinement in humans. The real power of such an approach can only now be fully realized through the development of advanced tools for monitoring immune response evolution at the single cell and molecular level. Here the ability to clone Ab genes from individual responding human B cells provides the opportunity to glean new insights into the specificity and functionality of evolving Ab repertoires, while next generation sequencing (NGS) approaches facilitate evolutionary study of responses at the clonotypic level. This project seeks to apply these tools to proof of concept (POC) studies aimed at demonstrating that DNA vaccination can provide a valuable tool to systematically probe evolving Ab repertoires in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 50 years on the day of screening
2. BMI between 18-30
3. Available for follow-up for the duration of the study
4. Willing and able to give written informed consent
5. At low risk of HIV infection and willing to remain so for the duration of the study defined as:

   * no history of injecting drug use in the previous ten years
   * no gonorrhoea or syphilis in the last six months
   * no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
   * no unprotected anal or vaginal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative
6. Willing to undergo HIV testing
7. Willing to undergo a genital infection screen, if indicated
8. If heterosexually active female, using an effective method of contraception with partner: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); bilateral tubual occlusion, vasectomised partner (if sole partner); sexual abstinence (based on historical preferred and usual lifestyle), from 30 days prior to the first vaccination until 30 days after the last, and willing to undergo urine pregnancy tests prior to each vaccination
9. If heterosexually active male, using male contraception (condom) with their partner from the first day of vaccination until 4 months after the last vaccination. Furthermore additional use of an effective method of contraception (as listed above) should be recommended for any non-pregnant female partner over the same period
10. Agree to abstain from donating blood for three months after the end of their participation in the trial, or longer if necessary
11. Registered with a GP for at least the past month
12. Entered and clearance obtained from The Overvolunteering Prevention System (TOPS)

Exclusion Criteria:

1. Pregnant or lactating
2. Use of any medical topical treatment on the injection or application site within the last four weeks
3. History of cardiac arrhythmia or palpitations (e.g, supraventricular tachycardia, atrial fibrillation, frequent ectopy), or sinus bradycardia prior to study entry (sinus arrhythmia is not excluded)
4. History of syncope or fainting episodes within 1 year of study entry
5. History of grand-mal epilepsy, seizure disorder or any history of prior seizure
6. Individuals in which a skin-fold measurement (cutaneous and subcutaneous tissue) of the upper right or left thigh exceeds 40 mm
7. Clinically relevant abnormality on history or examination
8. Known hypersensitivity to any component of the vaccine formulations used in this trial, or have severe or multiple allergies to drugs or pharmaceutical agents
9. History of severe local or general reaction to vaccination defined as

   * local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
   * general: fever ≥39.5°C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
10. Receipt of live attenuated vaccine within 30 days or other vaccine within 14 days of enrolment
11. Receipt of an experimental vaccine containing HIV antigens at any time in the past
12. Receipt of blood products or immunoglobin within 4 months of screening
13. Participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
14. HIV 1 or 2 positive or indeterminate on screening
15. Positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
16. Grade 1 or above routine laboratory parameters. Hyperbilirubinaemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia
17. Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators
18. Presence of any surgical or traumatic metal implants at the sites of administration
19. Unable to read and/or speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent
20. Unlikely to comply with protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | 12 Months
  Proportion of volunteers with moderate or greater reactogenicity (i.e., solicited adverse events) during a 7 day follow-up period after each vaccination.
vaccine-related unsolicited adverse events | 14 Months
  Proportion of volunteers with moderate or greater and/or vaccine-related unsolicited adverse events (AEs), including safety laboratory (biochemical, haematological) parameters, up to 28 days post each vaccination.
vaccine-related serious adverse events | 16 Months
  Proportion of volunteers with vaccine-related serious adverse events (SAEs) throughout the study period.

SECONDARY OUTCOMES:
Safety - event that occurred after vaccination | 12 Months
  Any grade of adverse event that occurs in a participant that has received at least one immunisation by either method.
Immunogenicity - kinetics of immune responses elicited by DNA vaccines | 12 Months
  To assess the kinetics of immune responses elicited by each of the DNA regimens:
  • Frequency and titer of serum binding antibodies to HIV CN54 gp140 antigen by ELISA.
Serum binding antibodies to HIV Env antigens | 12 Months
  Frequency, titer and avidity of serum binding antibodies to other HIV Env antigens (alternative clades) by ELISA or other assays.
Frequency and magnitude of HIV-gp140 specific B-cells | 12 Months
  Frequency and magnitude of HIV-gp140 specific B-cell-mediated responses in the systemic compartment measured by B-cell ELISPOT.
Mapping of serum binding antibodies | 12 Months
  Mapping of serum binding antibodies using Env subunit constructs (e.g., V2 scaffolds and hotspots) by ELISA.
Frequency and titer of serum neutralising antibodies | 12 Months
  Frequency and titer of serum neutralising antibodies to homologous virus, and, if warranted a wider a panel of viruses representing different clades.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fox, MD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Yes
Any publications based on the results of the Clinical Trial and originating from IC or the Investigators will be submitted for review to Ichor Medical Systems, Profectus Biosciences , UK HIV Vaccine Consortium (UK HVC) and Bill and Melinda Gates Foundation (BMGF), and will require their acceptance for further publications, according to the DNAVAC agreement
Supporting Information: CSR
Time Frame: 18 Months from when the clinical trial officially closed
Access Criteria: Directly from the PI of the clinical trial